CLINICAL TRIAL: NCT04001855
Title: Evaluating the Effect of Bathing Additives in Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left university
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1906687954
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: Randomized control split body study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dilute vinegar vs. dilute bleach bath (Experimental): Subjects will complete a total of 5 study visits over 11 days. At visits 1-4, subjects will soak their forearms in either dilute bleach or dilute vinegar for 10 minutes. At all visits, measurements of skin barrier function will be obtained using non-invasive, commercially-available devices. Non-invasive, non-painful tape stripping samples and skin culture swabs will also be collected.
  Interventions: Other: Dilute vinegar (acetic acid); Other: Dilute bleach
- Dilute vinegar vs. dilute bleach gauze soaks (Experimental): Subjects will complete a total of two study visits over 21 days, and will be instructed to apply gauze soaks daily at home over the 21-day study period. At baseline and 21-day follow-up visits, measurements of skin barrier function will be obtained using non-invasive, commercially-available devices. Non-invasive, non-painful tape stripping samples and skin culture swabs will also be collected. Subjects will also be provided with a non-invasive skin barrier measurement device to take daily recordings at home.
  Interventions: Other: Dilute vinegar (acetic acid); Other: Dilute bleach

INTERVENTIONS:
Other: Dilute vinegar (acetic acid) — Dilute vinegar baths or gauze soaks
Other: Dilute bleach — Dilute bleach baths or gauze soaks

SUMMARY:
This proposed project will be an open-label, split-arm, randomized controlled pilot study. Up to 60 patients diagnosed with atopic dermatitis (eczema) will be enrolled in the study. The purpose of this study is to understand the change in skin barrier function and skin microbial composition in patients with atopic dermatitis following dilute bleach bath/soak and dilute vinegar bath/soak.

DETAILED DESCRIPTION:
Atopic dermatitis (AD), also known as eczema, is an inflammatory skin condition that affects children and adults and causes skin redness, dryness and itching. Dilute bleach baths are standard of care for treatment of AD and work to decrease skin inflammation and modulate the skin microbiome. Dilute vinegar (acetic acid) has been reported to have similar effects on the skin. The purpose of this study is to evaluate the change in skin barrier function and skin microbial composition following baths or gauze soaks with dilute bleach and dilute vinegar.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, at least 5 years of age
* Subjects, parents/legal guardians must be able to comprehend and read the English language
* Subjects must have a diagnosis of atopic dermatitis (AD) by a board-certified dermatologist

Exclusion Criteria:

* Subjects who do not fit the inclusion criteria
* Subjects unable or unwilling to comply with the study procedures
* Concurrently have other inflammatory skin conditions
* Prior known allergies to any components of the materials used
* A subject who in the opinion of the investigator will be uncooperative or unable to comply with study procedures
* Subject unable to speak or read the English language
* Those that are pregnant, prisoners or cognitively impaired

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Skin barrier function - Transepidermal water loss (TEWL) | Up to 21 days
  Assess skin barrier function through measurement of transepidermal water loss (in g/m^2h) using a commercially-available, non-invasive device (Delfin VapoMeter: http://www.delfintech.com/en/product_information/vapometer/).
Skin barrier function - Stratum corneum hydration | Up to 21 days
  Assess skin barrier function through measurement of stratum corneum hydration (in arbitrary units) using a commercially-available, non-invasive device (Delfin MoistureMeterSC: http://www.delfintech.com/en/product_information/moisturemetersc/).
Skin barrier function - pH | Up to 21 days
  Assess skin barrier function through measurement of stratum corneum pH (in pH units) using a commercially-available, non-invasive device.
Skin culture swab | Up to 21 days
  Assess microbial composition via collection of non-invasive, non-painful skin culture swab samples.
Change in Eczema Area and Severity Index (EASI) | Up to 21 days.
  Clinical grading of atopic dermatitis/eczema severity (higher EASI scores indicating more severe AD).

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medicine Dermatology, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No